CLINICAL TRIAL: NCT03669900
Title: Radiological Measurements in Patients With Mild to Severe Hallux Valgus After Correction Surgery (SERI)
Brief Title: Outcomes of Hallux Valgus Correction Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Security Forces Hospital (Other)
Responsible Party: Principal Investigator, Raheef Alatassi, Orthopedic Surgeon, Security Forces Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hallux Valgus and SERI
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Hallux Valgus
Keywords: SERI; correction surgery; Complications; radiological; outcomes
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a minimally invasive surgery (SERI) (Other): The surgery consisted of varus traction, skin incision, metatarsal osteotomy and K- wire insertion. All the cases were done by the senior consultant orthopedic surgeon, including preoperative planning, the osteotomy itself and the follow up in the clinic. Another orthopedic surgeon was involved in collecting the data, doing all the measurements preoperative and postoperative and assisting the primary surgeon during the surgery.
  Interventions: Procedure: a minimally invasive surgery (SERI)

INTERVENTIONS:
Procedure: a minimally invasive surgery (SERI) — The SERI technique (as abbreviated to stand for simple, effective, rapid and inexpensive) was presented by several authors to be a minimally invasive technique since it presents with the same advantages as the percutaneous techniques with less tissue dissection and a need for only temporary hardware, meaning no instrumentation and surgery is performed under direct vision without fluoroscopy

SUMMARY:
HV correction surgery using SERI appear to sufficiently reduce the severity of HV deformity in all radiological measurements (HVA, IMA, DMAA) and the correction of subluxation of the first MTP joint and the sesamoids. SERI technique is an easy, inexpensive, less invasive, more cosmetic, with shorter operative time and with minimal complication rates.

To our knowledge, there is no report regarding HV treatment using SERI from Saudi Arabia or in any part of the Middle East. Therefore, this study conducted to determine the radiological measurements done preoperatively and compare the measurements done at one year postoperatively, recording the complication happened and measuring the cost effectiveness of such procedure.

DETAILED DESCRIPTION:
Hallux valgus (HV) is defined as a complex deformity where there is a lateral deviation of the proximal phalanx on the first metatarsal head (hallux) that is frequently associated with medial deviation of the first metatarsal, which may sometimes be accompanied by a significant functional disability and foot pain. Worldwide estimates from reports show a prevalence of 23% among adults below 65 years old and 35.7% among adults >65 years old, higher among females, and directly proportional to increasing age.

Because of the concomitant pain and other functional disability with HV, surgery is indicated usually depending on the degree of deformity based on the radiological findings as well as the physical examination findings. Radiological assessment includes weight-bearing anteroposterior (AP) and lateral imaging of the foot. The severity of the deformity is usually classified as mild, when the hallux valgus angle (HVA) is up to 19o , intermetatarsal angle (IMA) up to 13o; moderate when HVA is 20o to 40o; and severe when HVA is >40o and IMA >20o.

There were a multitude of modern concepts in the surgical treatment of HV, including the Keller's procedure, the distal soft-tissue procedure, osteotomies of the first metatarsal, distal metatarsal osteotomies (Wilson procedure, Mitchell osteotomy, distal Chevron osteotomy), and many other type of surgeries including diaphyseal osteotomies and arthrodesis. Most of these surgical procedures were shown to provide morphologic and functional re-balance after surgery. While there are more than 150 surgical procedures described to treat HV, none of them is considered as a gold standard and each one had it is own advantages and disadvantages.

Minimally invasive techniques for correction of HV include arthroscopy, percutaneous and minimum incision surgery which were found to provide better outcome by decreasing recovery and rehabilitation time. On the other hand, some authors suggested that to correct HV deformity using SERI, a lateral soft tissue release should be performed first and reposition the sesamoids to avoid recurrence of the HV.

The SERI technique (as abbreviated to stand for simple, effective, rapid and inexpensive) was presented by several authors to be a minimally invasive technique since it presents with the same advantages as the percutaneous techniques with less tissue dissection and a need for only temporary hardware, meaning no instrumentation and surgery is performed under direct vision without fluoroscopy. It is a type of distal first metatarsal osteotomy. Several studies using SERI have shown adequate correction of the deformity without avascular necrosis of the metatarsal head, pseudoarthrosis or recurrence.

Radiographic assessment including angular radiological parameters, sesamoid subluxation, and the articular congruency were shown to prove adequate correction of angular HV deformities. Preoperatively, measuring the axial view of the sesamoid position in the radiographic assessment of HV was proven to guide the surgeon on the appropriate surgical technique. Furthermore, measurements of the HVA and the IMA were recommended to evaluate preoperative assessment of the severity of HV and postoperative outcome of surgical treatment of HV.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged 20 years old to 60 years old admitted and managed for hallux valgus during the last 3 years (2013 - 2016) at Security Forces Hospital, Riyadh, Saudi Arabia.
* Reducible mild or moderate HV, HVA of ≤40o, IMA ≤20o with some severe cases.
* Patient with arthritis of the 1st MTP joint up to grade 2 according to the Regnauld's classification
* At least 2 years of follow-up in the hospital.

Exclusion Criteria:

* Patients who have stiffness of the first MTP joint
* Patients with severe arthritis of the first MTP joint (more than Regnauld's grade 2)
* Patients with history of rheumatoid arthritis or other inflammatory diseases, diabetics.
* Patients with neurological disorders.
* Patients with prior hallux surgery.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-25 (Actual)

PRIMARY OUTCOMES:
radiological measurements | one year
  Radiological assessment includes weight-bearing anteroposterior (AP) and lateral imaging of the foot. The severity of the deformity is usually classified as mild, when the hallux valgus angle (HVA) is up to 19o , intermetatarsal angle (IMA) up to 13o; moderate when HVA is 20o to 40o; and severe when HVA is >40o and IMA >20o

CONTACTS AND LOCATIONS:
Overall Officials: Talal Almalki, FRCS, Study Director — Security Forces Hospital
Locations (1):
- Security Forces Hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Nix S, Smith M, Vicenzino B. Prevalence of hallux valgus in the general population: a systematic review and meta-analysis. J Foot Ankle Res. 2010 Sep 27;3:21. doi: 10.1186/1757-1146-3-21. PMID 20868524
- [Background] Roddy E, Zhang W, Doherty M. Prevalence and associations of hallux valgus in a primary care population. Arthritis Rheum. 2008 Jun 15;59(6):857-62. doi: 10.1002/art.23709. PMID 18512715
- [Background] Robinson AH, Limbers JP. Modern concepts in the treatment of hallux valgus. J Bone Joint Surg Br. 2005 Aug;87(8):1038-45. doi: 10.1302/0301-620X.87B8.16467. No abstract available. PMID 16049235
- [Background] Giannini S, Cavallo M, Faldini C, Luciani D, Vannini F. The SERI distal metatarsal osteotomy and Scarf osteotomy provide similar correction of hallux valgus. Clin Orthop Relat Res. 2013 Jul;471(7):2305-11. doi: 10.1007/s11999-013-2912-z. Epub 2013 Mar 14. PMID 23494184
- [Background] Maffulli N, Longo UG, Marinozzi A, Denaro V. Hallux valgus: effectiveness and safety of minimally invasive surgery. A systematic review. Br Med Bull. 2011;97:149-67. doi: 10.1093/bmb/ldq027. Epub 2010 Aug 14. PMID 20710024
- [Background] Wu GB, Yang YF, Yu GR, Li B. Comment on Giannini et al.: A minimally invasive technique for surgical treatment of hallux valgus: simple, effective, rapid, inexpensive (SERI). Int Orthop. 2014 Mar;38(3):671-2. doi: 10.1007/s00264-013-2209-6. Epub 2013 Dec 5. No abstract available. PMID 24326360
- [Background] Giannini S, Faldini C, Nanni M, Di Martino A, Luciani D, Vannini F. A minimally invasive technique for surgical treatment of hallux valgus: simple, effective, rapid, inexpensive (SERI). Int Orthop. 2013 Sep;37(9):1805-13. doi: 10.1007/s00264-013-1980-8. Epub 2013 Jul 3. PMID 23820757
- [Background] Wagner E, Ortiz C, Torres K, Contesse I, Vela O, Zanolli D. Cost effectiveness of different techniques in hallux valgus surgery. Foot Ankle Surg. 2016 Dec;22(4):259-264. doi: 10.1016/j.fas.2015.11.004. Epub 2015 Dec 2. PMID 27810025
- [Background] Trnka HJ, Krenn S, Schuh R. Minimally invasive hallux valgus surgery: a critical review of the evidence. Int Orthop. 2013 Sep;37(9):1731-5. doi: 10.1007/s00264-013-2077-0. Epub 2013 Aug 29. PMID 23989262
- [Background] Lin YC, Cheng YM, Chang JK, Chen CH, Huang PJ. Minimally invasive distal metatarsal osteotomy for mild-to-moderate hallux valgus deformity. Kaohsiung J Med Sci. 2009 Aug;25(8):431-7. doi: 10.1016/S1607-551X(09)70538-8. PMID 19605337
- [Background] Thordarson D, Ebramzadeh E, Moorthy M, Lee J, Rudicel S. Correlation of hallux valgus surgical outcome with AOFAS forefoot score and radiological parameters. Foot Ankle Int. 2005 Feb;26(2):122-7. doi: 10.1177/107110070502600202. PMID 15737253
- [Background] Nery C, Coughlin MJ, Baumfeld D, Ballerini FJ, Kobata S. Hallux valgus in males--part 2: radiographic assessment of surgical treatment. Foot Ankle Int. 2013 May;34(5):636-44. doi: 10.1177/1071100713475351. Epub 2013 Jan 30. PMID 23637233
- [Background] Catanese D, Popowitz D, Gladstein AZ. Measuring sesamoid position in hallux valgus: when is the sesamoid axial view necessary? Foot Ankle Spec. 2014 Dec;7(6):457-9. doi: 10.1177/1938640014539804. Epub 2014 Jul 7. PMID 25005702
- [Background] Shima H, Okuda R, Yasuda T, Jotoku T, Kitano N, Kinoshita M. Radiographic measurements in patients with hallux valgus before and after proximal crescentic osteotomy. J Bone Joint Surg Am. 2009 Jun;91(6):1369-76. doi: 10.2106/JBJS.H.00483. PMID 19487514
- [Background] Coughlin MJ, Freund E. Roger A. Mann Award . The reliability of angular measurements in hallux valgus deformities. Foot Ankle Int. 2001 May;22(5):369-79. doi: 10.1177/107110070102200503. PMID 11428754
- [Derived] Almalki T, Alatassi R, Alajlan A, Alghamdi K, Abdulaal A. Assessment of the efficacy of SERI osteotomy for hallux valgus correction. J Orthop Surg Res. 2019 Jan 24;14(1):28. doi: 10.1186/s13018-019-1067-3. PMID 30678713